CLINICAL TRIAL: NCT00767754
Title: Phase 4 Study of Panic Disorder That Expresses to Change of Cerebral Glucose Metabolism After 12 Week of Paroxetine Treatment
Brief Title: Changes of Cerebral Glucose Metabolism After 12 Weeks of Paroxetine Treatment in Panic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Bum-Hee Yu, M.D. Ph.D. / Professor, Department of Psychiatry, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC IRB 2006-07-091; NCT00515749 (obsolete NCT alias)
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Panic Disorder
Keywords: panic disorder; paroxetine; PET
MeSH Terms: conditions — Panic Disorder | interventions — Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- paroxetine cr (Other): single arm
  Interventions: Drug: Paxil CR

INTERVENTIONS:
Drug: Paxil CR — 12 week treatment of Paxil(20-40mg)

SUMMARY:
Panic disorder is one of the most prevalent and disabling psychiatric disorders. Brain regions such as amygdala, hippocampus, periaqueductal gray (PAG), locus coeruleus, parahippocampal gyrus, frontal cortex, and thalamus has been reported to be related with the pathophysiology and treatment outcome in panic disorder. Paroxetine has been used as primary agent for treatment of panic disorder but there is little information on how paroxetine affects the brain function in patients with panic disorder.

The specific aim of this study is to examine the differences in brain activity between responders and nonresponders and to determine the predictor of paroxetine treatment in patients with panic disorder in terms of brain activity.

ELIGIBILITY:
Inclusion Criteria:

* panic disorder 20-60 years

Exclusion Criteria:

* history of major psychosis (schizophrenia or bipolar disorder), social phobia, obsessive-compulsive disorder, and generalized anxiety disorder, and posttraumatic stress disorder, alcohol abuse and dependence, current regular use of benzodiazepines
* less than 17 on the HAM-D

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2007-01; Primary Completion 2007-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
18FDG PET, PDSS & HAM-A | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bum-Hee Yu, M.D., Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea